CLINICAL TRIAL: NCT02448316
Title: Randomized Clinical Trial Comparing Conventional Conservative Treatment for Plantar Fasciopathia With Endoscopic Surgery With Fascial Release.
Brief Title: Plantar Fasciitis, Operation or Conservative Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Finn Elkjær Johannsen, chief physician, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2012-151
Record Dates: First submitted 2015-05-10; First posted 2015-05-19 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2017-03

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Endoscopy; Methylprednisolone; Methylprednisolone Acetate; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endoscopic surgery (Active Comparator): Endoscopic operation through 2 portals profound for the fascia plantaris
  Interventions: Procedure: endoscopic surgery
- conservative treatment (Active Comparator): The standard treatment here acting as controle treatment . All patients are informed to decrease activity level, use shoes with good shock absorption and are recommended to use insoles (standard orthoses) for increased shock absorption. Training is supervised every third week by a physiotherapist (week 1,3,6,9), and daily training is carried out at home. Glucocorticoid injections of 1 ml Glucocorticosteroid (methylprednisolon 40 mg) and 1 ml of Lidokaine 5mg/ml from the medial side profound to the thickened part of the fascia plantaris are given every month until the fascia thickness is below 4 mm (max 3 injections).
  Interventions: Drug: methylprednisolon; Drug: lidokaine; Behavioral: Training

INTERVENTIONS:
Procedure: endoscopic surgery — Through 2 portals profound for the fascia plantaris (deep-fascial) lateral and medial a heel-spur will be resected and the medial half of the fascia is released from its attachment to the calcaneus.
  A mikroskopic X-ray sensitive pearle (Tantalum-pearle) will be inserted in the fascia in the proximal end of the distal part of the remaining fascia for measuring distance (resorbtion).
  Three weeks after operation, the patients are instructed to start a specific training program. Training is supervised every third week by a physiotherapist (week 3,6,9,12 after operation), and daily training is carried out at home. Sutures are removed after 10 days,
  Other Names: Fascial release; Heel spur resection; Training
  Arms: endoscopic surgery
Drug: methylprednisolon — 1ml methylprednisolon is mixed with 1ml of Lidocain and injected underneath the plantar fascia as close to the medial attachment on calcaneus as possible
  Other Names: Depo-medrol; Glucocorticosteroid injection
  Arms: conservative treatment
Drug: lidokaine — 1ml methylprednisolon is mixed with 1ml of Lidocain and injected underneath the plantar fascia as close to the medial attachment on calcaneus as possible
  Other Names: Xylocain
  Arms: conservative treatment
Behavioral: Training — the patient is instructed in reduction in impact. strength training 3 times weekly and stretching exercises daily are recommended.
  Other Names: strength training; stretching
  Arms: conservative treatment

SUMMARY:
The purpose of this study is to compare in a randomized controlled trial the effect of endoscopic operation with the standard conservative treatmentprotocol with training supplemented with 1-3 injections of glucocorticoids in patients with chronic plantar fasciopathia.

DETAILED DESCRIPTION:
Plantars fasciitis (PF) is a frequently diagnosed condition, defined as pain at the medial tubercle of the calcaneus, and 10% of the population will at some points in their life experience this condition. Accumulated loading of the plantar fascia seems to relate to development of PF, as it is commonly seen in runners and those who are overweight, and number of daily steps or simply time of standing has been shown to be a predisposing factor for PF development ( Orthosis and glucocorticoid injections are 2 widely used treatments and in most clinics the standard treatment, despite the fact that a recent Cochrane review found limited evidence for treatment of plantar heelpain.

Once the condition gets chronic the response to several kinds of treatment is less predictable. However it has been demonstrated that endoscopic surgery for plantar fasciitis using a deep-fascial approach was successful in individuals with an active sports anamnesis, and all patients returned with this treatment to full athletic activities within 8-15 weeks. This high succesrate is not seen in conservative treatment with decrease in activity, training and injections of glucocorticosteroid, eventhough they had shorter disease duration. Therefore the investigators think it would be interesting to offer this minimal invasive operation to patients much earlier in the disease, especially as there is no reported severe sideeffects .

However, surgery is very seldom compared with results of other treatment modalities, and no randomized studies exist on the effect of operation vs the normal conservative standard-treatment.

The purpose of this study is to compare in a randomized controlled trial the effect of endoscopic operation with the standard conservative treatmentprotocol with training supplemented with 1-3 injections of glucocorticoids in patients with chronic plantar fasciopathia.

ELIGIBILITY:
Inclusion Criteria:

* pain at the medial attachment of fascia plantaris
* first step pain in the morning
* symptoms for at least 3 months
* ultrasound scanning at the first visit shows thickness of the proximal fascia above 4 mm
* patient can read and understand danish

Exclusion Criteria:

* known arthritis inflammatory bowl disease, psoriasis or clinical signs of any of these.
* leg ulcerations
* long lasting oedema of the leg and foot
* palpatory decreased puls in the foot
* diabetes
* reduced sensibility in the foot
* infections in the foot
* daily use of pain killers
* pregnancy or planning to become pregnant
* earlier operations on the foot, that is judged to complicate training.
* patients assessed not to be able to participate in the training for other reasons
* Glucocorticosteroid injection to the diseased plantar fascia within the last 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Foot Function Index | 6 months
  Foot Function Index (FFI) is a validated score usefull for plantar fasciitis. It consists of 23 questions concerning pain, function and impact on daily life. Each question is answered on a box scale 0-10, giving a score range: 0-230
Foot Function Index | 12 months
  Foot Function Index (FFI) is a validated score usefull for plantar fasciitis. It consists of 23 questions concerning pain, function and impact on daily life. Each question is answered on a box scale 0-10, giving a score range: 0-230

SECONDARY OUTCOMES:
100 mm VAS score for morning pain | 3 months
100 mm VAS score for morning pain | 6 months
100 mm VAS score for morning pain | 12 months
100 mm VAS score for morning pain | 24 months
100 mm VAS score for pain at function | 3 months
100 mm VAS score for pain at function | 6 months
100 mm VAS score for pain at function | 12 months
100 mm VAS score for pain at function | 24 months
single leg jumping length | 12 months
  Standing on the diseased leg, the patient jumps as far as possible landing on the same leg. the best of 3 trials.
positionel MR scanning (pMRI) | 12 months
  only for the operated patients the change in bone position in standing is measured using a pMRI, where bone position is measured in supine and standing before and 12 months after the operation. This will also include patients referred directly to operation and therefore not included in the RCT
Tantalum pearle-calcaneus distance | 12 months
  only for operated patients the distance from calcaneus to a Tantalum pearle inserted in the plantar fascia during operation is measured by lying and standing X-ray. This will also include patients referred directly to operation and therefore not included in the RCT
Foot Function Index | 24 months
  Foot Function Index (FFI) is a validated score usefull for plantar fasciitis. It consists of 23 questions concerning pain, function and impact on daily life. Each question is answered on a box scale 0-10, giving a score range: 0-230

CONTACTS AND LOCATIONS:
Overall Officials: Finn MD Johannsen, MD, Principal Investigator — Institute of Sports Medicine Copenhagen, Bispebjerg Hospital Copenhagen, Denmark
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Baldassin V, Gomes CR, Beraldo PS. Effectiveness of prefabricated and customized foot orthoses made from low-cost foam for noncomplicated plantar fasciitis: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Apr;90(4):701-6. doi: 10.1016/j.apmr.2008.11.002. PMID 19345789
- [Background] Crawford F, Thomson C. Interventions for treating plantar heel pain. Cochrane Database Syst Rev. 2003;(3):CD000416. doi: 10.1002/14651858.CD000416. PMID 12917892
- [Background] Neufeld SK, Cerrato R. Plantar fasciitis: evaluation and treatment. J Am Acad Orthop Surg. 2008 Jun;16(6):338-46. doi: 10.5435/00124635-200806000-00006. PMID 18524985
- [Background] Tsai WC, Hsu CC, Chen CP, Chen MJ, Yu TY, Chen YJ. Plantar fasciitis treated with local steroid injection: comparison between sonographic and palpation guidance. J Clin Ultrasound. 2006 Jan;34(1):12-6. doi: 10.1002/jcu.20177. PMID 16353228
- [Background] Uden H, Boesch E, Kumar S. Plantar fasciitis - to jab or to support? A systematic review of the current best evidence. J Multidiscip Healthc. 2011;4:155-64. doi: 10.2147/JMDH.S20053. Epub 2011 May 24. PMID 21655342
- [Background] Komatsu F, Takao M, Innami K, Miyamoto W, Matsushita T. Endoscopic surgery for plantar fasciitis: application of a deep-fascial approach. Arthroscopy. 2011 Aug;27(8):1105-9. doi: 10.1016/j.arthro.2011.02.037. Epub 2011 Jun 24. PMID 21704466
- [Background] Bazaz R, Ferkel RD. Results of endoscopic plantar fascia release. Foot Ankle Int. 2007 May;28(5):549-56. doi: 10.3113/FAI.2007.0549. PMID 17559761
- [Background] Jerosch J, Schunck J, Liebsch D, Filler T. Indication, surgical technique and results of endoscopic fascial release in plantar fasciitis (E FRPF). Knee Surg Sports Traumatol Arthrosc. 2004 Sep;12(5):471-7. doi: 10.1007/s00167-004-0496-6. Epub 2004 Apr 14. PMID 15088083
- [Background] Kalaci A, Cakici H, Hapa O, Yanat AN, Dogramaci Y, Sevinc TT. Treatment of plantar fasciitis using four different local injection modalities: a randomized prospective clinical trial. J Am Podiatr Med Assoc. 2009 Mar-Apr;99(2):108-13. doi: 10.7547/0980108. PMID 19299346